CLINICAL TRIAL: NCT06044051
Title: Dynamique Des Microbiomes Respiratoires Des Voies supérieures et inférieures associée à l'Asthme sévère Des Nourrissons
Brief Title: Dynamics of the Upper and Lower Airway Respiratory Microbiomes Associated With Severe Infant Asthma
Acronym: Microbiosthme
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023/0091/OB
Record Dates: First submitted 2023-07-27; First posted 2023-09-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Asthma in Children; Asthma
Keywords: microbiosme; Asthma in infant
MeSH Terms: conditions — Asthma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): All patients included will be followed for 1 year, every 3 months
  Interventions: Other: Blood sample; Other: Expectoration; Other: Nasopharyngeal swab

INTERVENTIONS:
Other: Blood sample — An additionnal volume of blood will be collected at inclusion and at each follow-up visit
Other: Expectoration — Expectoration will be collected at inclusion and at each follow-up visit
Other: Nasopharyngeal swab — A nasopharyngeal swab will be collected at inclusion and at each follow-up visit after an induced sputum

SUMMARY:
Nature of potential dysbiosis, interrelation of the different microbiomes of the respiratory tract, and potential role of the immune system in the pathogenesis of severe asthma in infants, and its evolution under treatment.

Exploring and understanding these data is to improve patient care and discover new therapeutic targets.

The aim is to open up prospects for therapeutic studies, such as the use of azithromycin as an immunomodulator in infant asthma, the results of which are discordant.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than 24 months old
* Follow-up by a pneumo-pediatrician for severe asthma in infants
* Requiring etiological investigations and assessment of severity in day hospitalization, including bronchial fibroscopy (HAS 2009)
* Parent informed of the research and having signed consent

Exclusion Criteria:

* Prematurity <32 WA
* Congenital heart disease with significant left to right shunt
* Chronic respiratory disease other than infant asthma (cystic fibrosis, bronchiolitis obliterans)
* Antibiotic therapy in progress or administered the seven days preceding the date of inclusion (day hospitalization)
* Refusal of bronchial fibroscopy

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2026-09-26 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
description of microbiomes from bronchoalveolar fluids | Inclusion
  analysis of bronchoalveolar fluids - NGS sequencing
description of microbiomes from nasopharyngeal samples | Inclusion
  analysis of nasopharyngeal samples- NGS sequencing
description of microbiomes from sputum samples | Inclusion
  analysis of sputum samples- NGS sequencing
description of microbiomes from bronchoalveolar fluids | at 3 months
  analysis of bronchoalveolar fluids- NGS sequencing
description of microbiomes from nasopharyngeal samples | at 3 months
  analysis of nasopharyngeal samples- NGS sequencing
description of microbiomes from sputum samples | at 3 months
  analysis of sputum samples- NGS sequencing
description of microbiomes from bronchoalveolar fluids | at 6 months
  analysis of bronchoalveolar fluids- NGS sequencing
description of microbiomes from nasopharyngeal samples | at 6 months
  analysis of nasopharyngeal samples- NGS sequencing
description of microbiomes from sputum samples | at 6 months
  analysis of sputum samples- NGS sequencing
description of microbiomes from bronchoalveolar fluids | at 9 months
  analysis of bronchoalveolar fluids - NGS sequencing
description of microbiomes from nasopharyngeal samples | at 9 months
  analysis of nasopharyngeal samples- NGS sequencing
description of microbiomes from sputum samples | at 9 months
  analysis of sputum samples- NGS sequencing
description of microbiomes from bronchoalveolar fluids | at 12 months
  analysis of bronchoalveolar fluids- NGS sequencing
description of microbiomes from nasopharyngeal samples | at 12 months
  analysis of nasopharyngeal samples- NGS sequencing
Description of microbiomes from sputum samples | at 12 months
  analysis of sputum samples- NGS sequencing

CONTACTS AND LOCATIONS:
Overall Officials: PETAT Hortense, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

REFERENCES:
- [Derived] Petat H, Hassel C, Michel A, Charbonnier C, Plantier JC, Marguet C. Microbiosthma: a prospective study following respiratory microbiota in young children with severe preschool wheezing to better understand their respiratory future. BMC Pulm Med. 2025 Jul 16;25(1):342. doi: 10.1186/s12890-025-03812-9. PMID 40670979